CLINICAL TRIAL: NCT01124890
Title: Southwest German Interventional Study in Acute Myocardial Infarction III
Acronym: SIAMIII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BS S3
Record Dates: First submitted 2010-05-11; First posted 2010-05-17 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; thrombolysis; percutaneous coronary interention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conservative (Placebo Comparator): no transfer for early percutaneous coronary intervention after thrombolysis
  Interventions: Device: late percutaneous coronary intervention
- early PCI (Active Comparator): transfer for early percutaneous coronary intervention after thrombolysis
  Interventions: Device: early percutaneous coronary intervention

INTERVENTIONS:
Device: early percutaneous coronary intervention
  Arms: early PCI
Device: late percutaneous coronary intervention
  Arms: Conservative

SUMMARY:
SIAM III was a multicenter, randomized, prospective, controlled trial in patients with ST-elevation myocardial infarction receiving fibrinolysis <12 hours after onset of symptoms. Patients of the early PCI group were transferred within 6 hours after fibrinolysis for PCI. The conservative group received elective PCI two weeks after fibrinolysis.

DETAILED DESCRIPTION:
SIAM III was a multicenter, randomized, prospective, controlled trial in patients with ST-elevation myocardial infarction receiving fibrinolysis <12 hours after onset of symptoms. All patients received reteplase, aspirin in combination with ticlopidin, and heparin. Patients of the early PCI group were transferred within 6 hours after fibrinolysis for PCI. The conservative group received elective PCI two weeks after fibrinolysis. In total 197 patients were included, 163 were treated by PCI. The primary end point was the composite of ischemic events, death, reinfarction, and target lesion revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of MI present for 12 h
* ST segment elevation of at least 1 mm in two or more limb leads,
* ST segment elevation of at least 2 mm in the precordial leads,
* or new bundlebranch block
* Patients eligible for thrombolysis
* Informed consent for participation

Exclusion Criteria:

* Secondary or iatrogenic infarction
* Chronic renal insufficiency requiring dialysis
* Coronary anatomy unsuitable for stent placement
* Anticipated indication for surgical coronary revascularization within 6 months
* Previous MI in the area of the infarct related vessel
* Infarct related lesion not clearly defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 1998-07; Primary Completion 2001-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 6 months
  The primary endpoint was a combined endpoint consisting of death, reinfarction, ischemic events, and target vessel revascularization.

SECONDARY OUTCOMES:
Death | 6 months
  Total mortality as well as cardiac and noncardiac deaths were counted.
Reinfarction | 6 months
  Reinfarction was defined as two or more of the following criteria: chest pain lasting for more than 30 minutes; a new significant ST-elevation; and a rise in the serum creatine kinase level to more than >3x upper normal limit.
Ischemic Events | 6 months
  Ischemic events included unplanned hospitalization and / or unplanned angiography due to postinfarction angina, recurrent angina pectoris lasting for more than 15 minutes despite the administration of nitrates, or being accompanied by electrocardiogram changes, pulmonary edema, or hypotension.
Target Vessel Revascularization | 6 months
  Target vessel revascularization was defined as any repeated percutaneous coronary intervention or coronary artery bypass graft surgery involving the infarct related lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, MD, Principal Investigator — University of Saarland
Locations (1):
- University Hospital, Klinik fuer Innere Medizin III, Homburg/Saar, Germany

REFERENCES:
- [Result] Scheller B, Hennen B, Hammer B, Walle J, Hofer C, Hilpert V, Winter H, Nickenig G, Bohm M; SIAM III Study Group. Beneficial effects of immediate stenting after thrombolysis in acute myocardial infarction. J Am Coll Cardiol. 2003 Aug 20;42(4):634-41. doi: 10.1016/s0735-1097(03)00763-0. PMID 12932593
- [Derived] Clever YP, Cremers B, Link A, Bohm M, Scheller B. Long-term follow-up of early versus delayed invasive approach after fibrinolysis in acute myocardial infarction. Circ Cardiovasc Interv. 2011 Aug;4(4):342-8. doi: 10.1161/CIRCINTERVENTIONS.111.962316. Epub 2011 Jun 28. PMID 21712524